CLINICAL TRIAL: NCT03641456
Title: Lenalidomide, Bortezomib, and Dexamethasone Combination Therapy as Induction Followed by Bortezomib and Lenalidomide Maintenance in Patients With Newly Diagnosed High Risk Multiple Myeloma
Brief Title: VRD as Induction Followed by VR Maintenance in Patients With Newly Diagnosed High Risk Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hua Wang, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-2018
Record Dates: First submitted 2018-08-11; First posted 2018-08-22 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Myeloma; Newly Diagnosed; High Risk
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Bortezomib; Lenalidomide; Dexamethasone; dexamethasone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VRD for Followed by VR (Experimental): The investigators gave patients subcutaneous bortezomib 1.3mg/m2 on days 1, 8,15, and 22; oral lenalidomide 25mg on days 1 to 21; and oral dexamethasone 40mg on days 1, 8, 15 and 12 of a 28-day cycle.Patients are allowed to proceed to stem-cell transplantation after four cycles of VRD at the discretion of the treating physician.Two months after hematologic recovery, nonprogressive patients are to receive consolidation therapy comprising two cycles of VRD.Patients who do not proceed to stem-cell transplantation receive more two induction cycles after obtaining maximum response but no less than six cycles totally. Responding patients could receive maintenance therapy comprising 4-week cycles of bortezomib 1.3mg/m2 on days 1 and 15 and lenalidomide on days 1 to 21 at the dose level of 10mg.
  Interventions: Drug: bortezomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: bortezomib — The investigators gave patients subcutaneous bortezomib 1.3mg/m2 on days 1, 8,15, and 22 of a 28-day cycle. More two induction cycles after obtaining maximum response but no less than six cycles totally.Responding patients could receive maintenance therapy comprising 4-week cycles of bortezomib on days 1 and 15 at the dose level of 1.3mg/m2. Patients discontinued treatment if they had progressive disease or or unacceptable toxic effects not controlled with dose modifications.
  Other Names: Velcade
Drug: Lenalidomide — The investigators gave patients oral lenalidomide 25mg on days 1 to 21 of a 28-day cycle. More two induction cycles after obtaining maximum response but no less than six cycles totally.Responding patients could receive maintenance therapy comprising 4-week cycles of lenalidomide on days 1 to 21 at the dose level of 10mg. Patients discontinued treatment if they had progressive disease or unacceptable toxic effects not controlled with dose modifications.
  Other Names: Revlimid
Drug: Dexamethasone — The investigators gave patients oral dexamethasone 40mg on days 1, 8, 15 and 22 of a 28-day cycle. More two induction cycles after obtaining maximum response but no less than six cycles totally.
  Other Names: Dexamethasone Acetate

SUMMARY:
The phase 2 study evaluated the efficacy and safety of bortezomib in combination with lenalidomide as maintenance therapy in high risk newly diagnosed multiple myeloma patients who receive lenalidomide,bortezomib, and dexamethasone Combination as induction therapy.

DETAILED DESCRIPTION:
The aim of front-line therapy for multiple myeloma (MM) is to substantially decrease tumor burden, either in preparation for consolidation with high-dose melphalan therapy with autologous stem cell transplantation (ASCT) or as a means in itself to provide long-term disease control. The degree of disease reduction is associated with improved outcome, including prolonged progression-free survival (PFS) and overall survival (OS),both after preparation for or after consolidation with ASCT,and in patients not proceeding to ASCT.The introduction of the proteasome inhibitor bortezomib and the immunomodulatory drugs thalidomide and lenalidomide has been associated with improved survival. Combinations of bortezomib or lenalidomide with conventional anti-MM drugs have demonstrated very high overall response rates and quality of response in the front-line setting, as reviewed recently.The phase 2 study evaluated the efficacy and safety of bortezomib in combination with lenalidomide as maintenance therapy in high risk newly diagnosed multiple myeloma patients who receive lenalidomide, bortezomib, and dexamethasone(VRD) Combination as induction therapy.The investigators gave patients subcutaneous bortezomib on days 1, 8,15, and 22; oral lenalidomide on days 1 to 21; and oral dexamethasone on days 1, 8, 15 and 12 of a 28-day cycle.Patients are allowed to interrupt therapy for collection of stem cells at any time after three cycles of induction, and to proceed to stem-cell transplantation after four cycles of induction at the discretion of the treating physician.Two months after hematologic recovery, nonprogressive patients are to receive consolidation therapy comprising two 4-week cycles of VRD or the second autologous hematopoietic stem cell transplantation (determined by the attending physician according to the patient's physical condition, willingness and the number of CD34 + cells collected).Patients who do not proceed to stem-cell transplantation receive a total of 12 courses of VRD induction therapy(dexamethasone dosage will be reduced to 20mg from the 9th course of treatment). Responding patients could receive maintenance therapy comprising 4-week cycles of bortezomib on days 1 and 15 at the dose level of 1.3mg/m2 and lenalidomide on days 1 to 21 at the dose level of 10mg.Participants discontinued treatment if participants had progressive disease or unacceptable toxic eff ects not controlled with dose modifications.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a newly diagnosis of multiple myeloma
* Patient requires treatment for multiple myeloma
* Subject have high-risk characteristics.Our definition for high risk multiple myeloma :(1) with cytogenetic abnormalities including del(17p),t(4;14),t(14;16),and/or t(14;20) ;(2) R-ISS III；(3) ISS III and no complete remission is achieved before maintenance therapy.
* Subject has measurable disease as defined by > 0.5 g/dL serum monoclonal protein, >10 mg/dL involved serum free light chain (either kappa or lambda) provided that the serum free light chain ratio is abnormal, >0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s) of at least 1cm in greatest dimension as measured by either CT scanning or MRI
* Subject has a Karnofsky performance status ≥60%
* Subject has a life expectancy ≥ 3 months
* Subjects must meet the following laboratory parameters:

Absolute neutrophil count (ANC) ≥750 cells/mm3 (1.0 x 109/L) Hemoglobin ≥ 7 g/dL Platelet count ≥ 75,000/mm3 (30 x 109/L if extensive bone marrow infiltration) Serum SGOT/AST <3.0 x upper limits of normal (ULN) Serum SGPT/ALT <3.0 x upper limits of normal (ULN) Serum total bilirubin <2.0 mg/dL (34 µmol/L) Creatinine clearance ≥ 30 cc/min

Exclusion Criteria:

* Subject has immeasurable MM (no measurable monoclonal protein, free light chains in blood or urine, or measureable plasmacytoma on radiologic scanning)
* Subject has a prior history of other malignancies unless disease-free for ≥ 5 years, except for basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or localized prostate cancer with Gleason score < 7 with stable prostate specific antigen (PSA) levels
* Subject has had myocardial infarction within 6 months prior to enrollment, or NYHA (New York Hospital Association) Class III or IV heart failure (see Appendix VI), Ejection Fraction < 35%, uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Female subject who is pregnant or lactating
* Subject has known HIV infection
* Subject has known active hepatitis B or hepatitis C infection
* Subject has active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program
* Subject is unable to reliably take oral medications
* Subject has a history of thromboembolic event within the past 4 weeks prior to enrollment
* Subject has any clinically significant medical or psychiatric disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Very good partial response or better by International Myeloma Working Group criteria | up to end of follow-up-phase (approximately 3 years)
  Number of participants with very good partial response or better as Assessed by International Myeloma Working Group criteria，change from baseline.

SECONDARY OUTCOMES:
progression free survival | up to end of follow-up-phase (approximately 3 years)
  Duration from start of the treatment to disease progression or death (regardless of cause of death), whichever comes first.
overall survival | up to end of follow-up-phase (approximately 3 years)
  Duration from start of the treatment to death (regardless of cause of death).
Incidence of Treatment-Emergent Adverse Events as Assessed by CTCAE v 4.0 | up to end of follow-up-phase (approximately 3 years)
  Number of participants with Treatment-Emergent Adverse Events as Assessed by CTCAE v 4.0，change from baseline
complete response rate by International Myeloma Working Group criteria | up to end of follow-up-phase (approximately 3 years)
  Number of participants with complete response as Assessed by International Myeloma Working Group criteria，change from baseline.
overall response rate by International Myeloma Working Group criteria | up to end of follow-up-phase (approximately 3 years)
  Number of participants with response (CR+VGPR+PR) as Assessed by International Myeloma Working Group criteria，change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Wang, MD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China